CLINICAL TRIAL: NCT06380296
Title: Clinical and Radiographic Outcomes of NeoMTA and NeoPUTTY Pulpotomies in Primary Molars: A Randomized Controlled Trial
Brief Title: Outcomes of NeoMTA and NeoPUTTY Pulpotomies in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Beatriz Ferraz dos Santos, Clinician-scientist; Research director, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-10240
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeoMTA (Active Comparator): Trained dentists will perform the primary molar pulpotomy following a standardized protocol. After amputation of the coronal pulp, the pulp chamber will be filled with NeoMTA 2. Tooth will be then restored with an appropriately sized stainless steel crown cemented with a glass ionomer cement at the same visit. Follow-up visits will be scheduled at 1, 6, 12 and 24 months after the procedure to assess the success rate of primary molars pulpotomy.
  Interventions: Other: Primary molars pulpotomies with NeoMTA
- NeoPUTTY (Experimental): Trained dentists will perform the primary molar pulpotomy following a standardized protocol. After amputation of the coronal pulp, the pulp chamber will be filled with NeoPUTTY. Tooth will be then restored with an appropriately sized stainless steel crown cemented with a glass ionomer cement at the same visit. Follow-up visits will be scheduled at 1, 6, 12 and 24 months after the procedure to assess the success rate of primary molars pulpotomy.
  Interventions: Other: Primary molar pulpotomies with NeoPUTTY

INTERVENTIONS:
Other: Primary molars pulpotomies with NeoMTA — Primary molar pulpotomies will be performed by trained dentists using NeoMTA, a bioactive material containing calcium silicate known for its bio-active and bone forming potential. Follow-up visits at 1, 6, 12 and 24 months will be conducted to assess success rate, and clinical and radiographic outcomes
  Arms: NeoMTA
Other: Primary molar pulpotomies with NeoPUTTY — Primary molar pulpotomies will be performed by trained dentists using NeoPUTTY, a ready to use bioactive material containing calcium silicate. Follow-up visits at 1, 6, 12 and 24 months will be conducted to assess success rate, and clinical and radiographic outcomes
  Arms: NeoPUTTY

SUMMARY:
The goal of this clinical trial is to evaluate the outcomes of different medications used for pulpotomies (baby root canal) in children. The main question it aims to answer is: • what are the long-term clinical and radiographic success of pulpotomies in baby teeth using two different medications (NeoMTA and NeoPUTTY) over a 24-month follow-up period? Healthy children aged between 3 and 10 years undergoing dental treatment under general anesthesia who have deep caries lesions approximating or reaching the nerve will be invited to participate in this study. Pulpotomies (baby root canal) will be performed by trained dentists following a protocol. Children will receive pulpotomies either with NeoMTA or NeoPUTTY, two medications indicated for the procedure. Participants will be asked to come for an appointment at 1, 6, 12 and 24 months after the procedure. Researcher will compare the clinical and radiographic performance of pulpotomies (baby root canal) done with both medications.

DETAILED DESCRIPTION:
This single-site, double-blinded (participants and evaluators) randomized clinical trial with parallel groups will be conducted at the Division of Dentistry, Montreal Children's Hospital. Healthy children aged between 3 and 10 years undergoing dental rehabilitation under general anesthesia who have deep caries lesions approximating or reaching the pulp without any signs or symptoms of pulpal degeneration in one or more primary molars will be invited to participate in this study. All participants will be randomly assigned (1:1 ratio) into two groups: i) pulpotomy with NeoMTA; and ii) pulpotomy with NeoPutty. Follow-up visits at 1, 6, 12 and 24 months will be conducted to assess the clinical and radiographic outcomes.

The sample size calculation was done using G*Power 3.1.9.4 software (Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany). In a recent study conducted by our research team, the 24-month success rates of NeoMTA pulpotomy in primary molars was 98% (manuscript in preparation for submission). To account for a desired accuracy of 20%, a significance level of 5%, and a safety margin of 20% to compensate for patient dropouts, a minimum sample size of 47 teeth in each group will be required.

Trained clinical staff f will perform all primary molar pulpotomies following a standardized protocol doe each pulp medication used (NeoMTA or NeoPUTTY).

A baseline questionnaire will be filled by caregivers to assess children's sociodemographic characteristics. At each follow-up visit, standardized clinical and radiographic will be performed by trained dentists.

The post-operative clinical success will be considered as a retained tooth that is void of signs and symptoms of infection such as pain on percussion, mobility, presence of a fistula, or an abscess. Radiographic success will be determined by the lack of pathologic changes such as internal or external root resorption, or a periradicular pathosis. The extraction of the tooth due to signs and symptoms of infection will be considered as a failure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 3 and 10 years
* Primary molars with no history of spontaneous or persistent pain
* Restorable primary molars with deep carious lesions approximating or reaching the pulp
* Primary molars with at least 2/3rd of the root length present
* Radiographically, the inclusion criteria were as follows: deep dentin caries approximating or reaching the pulp; no more than one-third of physiologic root resorption; no widening of the periodontal ligament (PDL) space; no pathologic internal or external root resorption; and no apical or furcal radiolucency.
* Children who can understand and speak French or English.

Exclusion Criteria:

* Primary molars with pathological mobility, tenderness to percussion, swelling, or sinus tract
* Primary molars without hemostasis after coronal pulp amputation within five minutes.
* Primary molars with widening of the periodontal ligament (PDL) space; pathologic internal or external root resorption; and apical or furcal radiolucency

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Success rate of a primary molar pulpotomy | 24 months
  A retained primary molar that is void of signs and symptoms of infection such as pain on percussion, mobility, presence of a fistula, or an abscess
Radiographic success of a primary molar pulpotomy | 24 months
  Absence of pathologic changes such as internal or external root resorption, or a periradicular pathosis.

IPD SHARING:
Plan to Share IPD: No